CLINICAL TRIAL: NCT05131451
Title: Autonomous AI for Diabetic Retinopathy Screening in Youth (AI-DR): A Randomized Control Trial
Brief Title: ACCESS: AI for pediatriC diabetiC Eye examS Study
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB00288043
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: 1. Control Arm - Standard of care referral to an eye care provider + Educational Reinforcement
  2. Intervention Arm - Point of Care Diabetic Retinopathy screening using Autonomous artificial intelligence on a non-mydriatic fundus camera
Masking Description: Participants are masked to the study arms until after randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Usual care with educational reinforcement (No Intervention): Standard of care referral to Eye Care Provider (ECP) for the diabetic eye exam with educational reinforcement
- Diabetic Retinopathy Exam (Experimental): Point of care (POC) Diabetic Retinopathy Exam using Autonomous AI on non-mydriatic fundus camera
  Interventions: Diagnostic Test: Point of Care Autonomous AI diabetic retinopathy exam

INTERVENTIONS:
Diagnostic Test: Point of Care Autonomous AI diabetic retinopathy exam — Participants will get a point of care diabetic retinopathy eye exam using autonomous AI. Those that test positive will be referred to Eye Care Provider for dilated eye exam.
  Other Names: IDx-DR
  Arms: Diabetic Retinopathy Exam

SUMMARY:
The purpose of this study is to determine if providing in clinic point-of-care autonomous AI diabetic retinopathy exams improves screening rates compared to standard of care referral to an eye care provider, in a randomized control trial in a racially and ethnically diverse cohort of youth.

DETAILED DESCRIPTION:
This study will recruit 164 individuals ages 8-21 with type 1 and type 2 diabetes. Participants will be randomized to usual care (referral to an eye care provider for a dilated eye exam) or the intervention arm and undergo a point-of-care diabetic eye exam using autonomous AI software on a non-mydriatic fundus camera. Participants in the intervention group will receive the diabetic eye exam results immediately from the autonomous AI system, and if abnormal will be referred to an eye care provider for a dilated eye exam. Participants in the standard of care group will have 6 months to complete the diabetic eye exam.

ELIGIBILITY:
Inclusion Criteria:

Meets American Diabetes Association (ADA) criteria for diabetic retinopathy screening:

* Diagnosis of Type 1 diabetes for ≥3 years, and age 11 or in puberty
* Diagnosis of Type 2 diabetes

Exclusion Criteria:

* Diabetic eye exam within the last 6 months
* Known diabetic retinopathy

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 164 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Risa Wolf, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Pediatric Diabetes Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetic Retinopathy Exam: Point of care (POC) Diabetic Retinopathy Exam using Autonomous AI (artificial intelligence) on non-mydriatic fundus camera
  Point of Care Autonomous AI diabetic retinopathy exam: Participants will get a point of care diabetic retinopathy eye exam using autonomous AI. Those that test positive will be referred to Eye Care Provider for dilated eye exam.
Period: Overall Study
Arm/Group | Usual Care With Educational Reinforcement | Diabetic Retinopathy Exam
Started | 83 | 81
Completed | 82 (One patient in the usual care arm was inadvertently enrolled in another eye screening study.) | 81
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care With Educational Reinforcement | Diabetic Retinopathy Exam | Total
Number analyzed (Participants) | 83 | 81 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (2.8) | 15.3 (2.8) | 15.2 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 49 | 96
  Male | 36 | 32 | 68
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 4 | 6 | 10
  Non-Hispanic Black | 32 | 26 | 58
  Hispanic | 5 | 5 | 10
  Non-Hispanic White | 42 | 44 | 86
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 83 | 81 | 164

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Get Screened With a Diabetic Eye Exam
Description: The number of participants who get screened with a diabetic eye exam will be assessed for the AI group and the standard of care group referral to an eye care provider (ECP).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care With Educational Reinforcement | Diabetic Retinopathy Exam
Number analyzed (Participants) | 82 | 81
Participants | 18 | 81

2. Secondary Outcome: Follow-up Rates With an Eye Care Provider
Description: The number of patients that follow-up with an eye care provider (ECP), for participants in the standard of care group referred to ECP, and for participants in the AI group with an abnormal exam result that are then referred to the ECP for a dilated eye exam.
Time Frame: 6 months
Population: The diabetic retinopathy exam group only includes those that had an abnormal AI exam and were referred to an eye care provider for a dilated eye exam.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care With Educational Reinforcement | Diabetic Retinopathy Exam
Number analyzed (Participants) | 82 | 25
Participants | 18 | 16

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Usual Care With Educational Reinforcement | Diabetic Retinopathy Exam
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/81
Other Adverse Events (participants affected / at risk) | 0/83 | 0/81

LIMITATIONS AND CAVEATS:
Autonomous AI is not FDA cleared for use in ages 21 and under. Some participants were familiar with autonomous AI diabetic eye exams from a prior study and may have been more accepting of participation in the current study.

Although pharmacologic dilation is not necessary in the pediatric population to obtain sufficient fundus imaging, this may not be applicable to adults where real-world studies have demonstrated higher rates of insufficient images without pharmacologic dilation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT05131451/Prot_SAP_000.pdf